CLINICAL TRIAL: NCT02240524
Title: A Phase III Study of Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Locally Advanced Gastric Cancer After radIcal Gastrectomy With D2 Lymphadenectomy
Brief Title: Efficacy of HIPEC in the Treatment of Patients With Locally Advanced Gastric Cancer
Acronym: HIPEC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014514
Record Dates: First submitted 2014-06-03; First posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Advanced Gastric Adenocarcinoma
Keywords: Gastric adenocarcinoma; HIPEC; Paclitaxel; Oxaliplatin; Capecitabine
MeSH Terms: interventions — Neoadjuvant Therapy; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D2 lymphadenectomy and HIPEC and Systemic chemotherapy (Experimental): Intraoperative and postoperative hyperthermic intraperitoneal chemotherapy (twice HIPEC) were performed after radical gastrectomy with D2 lymphadenectomy, followed by 8 cycles of systemic chemotherapy.
  HIPEC was conducted within 48 h after surgery: Normal saline 3000ml-4000ml, Paclitaxel 75mg/m^2, 43°C, 60min.
  Systemic chemotherapy (XELOX):
  Oxaliplatin: 130mg/m^2, d1, Intravenous infusion, every 3 weeks. Capecitabine: 1g/m^2 bid, days 1-14, every 3 weeks and maximum 8 cycles, or progression/intolerance.
  Interventions: Procedure: D2 lymphadenectomy; Procedure: Systemic chemotherapy; Procedure: HIPEC
- D2 lymphadenectomy+Systemic chemotherapy (Placebo Comparator): 8 cycles of systemic chemotherapy were performed after radical gastrectomy with D2 lymphadenectomy.
  Systemic chemotherapy (XELOX):
  Oxaliplatin: 130mg/m^2, d1, Intravenous infusion, every 3 weeks. Capecitabine: 1g/m^2 bid, days 1-14, every 3 weeks and maximum 8 cycles, or progression/intolerance.
  Interventions: Procedure: D2 lymphadenectomy; Procedure: Systemic chemotherapy

INTERVENTIONS:
Procedure: D2 lymphadenectomy — The dissected lymph nodes were classified according to the Japanese Classification of Gastric Carcinoma, first English edition.
Procedure: Systemic chemotherapy
Procedure: HIPEC
  Other Names: hyperthermic intraperitoneal chemoperfusion
  Arms: D2 lymphadenectomy and HIPEC and Systemic chemotherapy

SUMMARY:
The purpose of this study is to study the efficacy of hyperthermic intraperitoneal chemotherapy in the treatment of patients with locally advanced gastric cancer after radical gastrectomy with D2 lymphadenectomy. It is a multicentric and randomised phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 < age ≤ 65 years old
* Male or Non pregnant female
* The Eastern Cooperative Oncology Group (ECOG) status ≤ 2
* Histologically diagnosed as T4 gastric adenocarcinoma (determined from data obtained by endoscopic ultrasound or CT scan)
* Have not received cytotoxic chemotherapy, radiotherapy or immunotherapy
* White blood cells > 4,000/mm3
* neutrophils ≥ 1,500/mm3
* platelets ≥ 100,000/mm3
* hemoglobin>9g/l
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) < or = 2.5 times upper limit of nominal (ULN)
* total bilirubin (TBIL) < 1.5 times ULN
* serum creatinine < 1 times ULN
* Having given written informed consent prior to any procedure related to the study

Exclusion Criteria:

* Existence of macroscopic peritoneal implants
* Prior malignant tumors with detectable signs of recurrence or distant metastasis
* Poorly controlled disease e.g. atrial fibrillation, stenocardia, cardiac insufficiency, persistent hypertension despite medicinal treatment, ejection fraction<50%
* Receiving other cytotoxic chemotherapy
* High grade of intra-abdominal adhesions
* Contraindication to any therapy contained in this regimen specific to the study Without given written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  From the date of surgery to the date of death or to the end of follow-up

SECONDARY OUTCOMES:
Recurrence-free survival | 5 years
  From the date of surgery to the date of recurrence or to the end of follow-up
Locoregional-free survival | 5 years
  From the date of surgery to the date of locoregional recurrence or to the end of follow-up
Hepatic metastases-free survival | 5 years
  From the date of surgery to the date of recurrence or to the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: shuzhong cui, Ph.D, Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Department of Abdominal Surgery (Section 2), Affiliated Tumor Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China